CLINICAL TRIAL: NCT00501358
Title: Assessment of Sleep Apnea Syndrome as a Risk Factor for Venous Thromboembolism
Brief Title: Sleep Apnea and Tromboembolic Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Collaborators: Fundacion Caubet-Cimera Islas Baleares (Other)
Other Study IDs: TEP-SAHS
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2007-07-16 (Estimated); Status verified 2007-07

CONDITIONS: Sleep Apnea Syndromes; Venous Thromboembolism
Keywords: SLEEP APNEA; venous thromboembolism; COAGULABILITY; COAGULATION FACTORS; HYPOXIA
MeSH Terms: conditions — Sleep Apnea Syndromes; Venous Thromboembolism; Hypoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
There is some evidence for a hypercoagulable state in sleep apnea-hipopnea syndrome (SAHS), which could play a role in the increased cardiovascular morbility and mortality. Respiratory alterations (hypoxia, hypoxia- reoxygenation) and sleep fragmentation that these patients suffer during the sleep may induce modifications in clotting-fibrinolisis factors that may be a risk factor for venous thromboembolism (VTE).

OBJECTIVES:To calculate and compare the prevalence of sleep apnea-hipopnea syndrome in patients with venous thromboembolism with a gender, aged and BMI matched control group. Assessment of the association between SAHS and other risk factors for VTE. To compare clotting- fibrinolisis patterns, sleep parameters, blood pressure and pulmonary arterial obstruction index in patients with SAHS and VTE and those ones without SAHS.

DETAILED DESCRIPTION:
DESIGN: Case-control study.

METHODS: 133 SAHS patients and 133 controls will be studied. The study includes:

a) medical history; b) anthropometric variables (weight, height, body mass index, Mallampati index); c) sleepiness tested by Epworth scale; d) London Chest Activity of Daily Living Scale; e) conventional polysomnography (PSG); f) testing: clotting-fibrinolisis factors (factor V, VII, VIII; C and S protein, plasminogen tissular activator (t-PA) and inhibitor of plasminogen activator (PAI-1); g) d-dimer and thrombin-antithrombin III complex; h) basic biochemical profile and hemograma; i) Pulmonary artery obstruction index.

ELIGIBILITY:
Inclusion Criteria:

* Case group:
* Pulmonary embolism diagnosed by CT Pulmonary Angiography.
* Control group:
* randomly selected from among patients in two primary health care centers in Mallorca without tromboembolic disease

Exclusion Criteria:

* Refusal to sign informed consent.
* Expected survival less than 12 months
* Long-term oxygen therapy
* Hospital admission in the previous two months.
* Familiar thrombophilia

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Alonso, MD, Principal Investigator — Sociedad Española de Neumología y Cirugía Torácica
Locations (1):
- Hospital Universitario Son Dureta, Palma de Mallorca, Balearic Islands, Spain